CLINICAL TRIAL: NCT02384616
Title: Impact of Intraoperative High Inspired OXygen Fraction on Pulmonary Function, Surgical Site Infection, Postoperative Nausea and Vomiting in PEDiatric Anesthesia, the OXPED Study
Brief Title: Hyperoxygenation in Anesthetized Children
Acronym: OXPED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walid HABRE (Other)
Responsible Party: Sponsor-Investigator, Walid HABRE, Associate Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CER 14-039
Record Dates: First submitted 2015-02-17; First posted 2015-03-10 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Hyperoxia
Keywords: Lung Volume Measurements; airway resistance; general anesthesia
MeSH Terms: conditions — Hyperoxia | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group High FiO2 (Active Comparator): Children will receive Fi02 100% during induction of anesthesia until end tidal oxygen concentration (Et 02) of 90% before intubation, anesthesia will be maintained with Fi02 of 80%. Then, shortly before the planned extubation, Fi02 will be increased to 100%.
  Interventions: Other: Oxygen
- Group Low FiO2 (Active Comparator): Children will receive Fi02 80% until Et 02 70% before intubation, anaesthesia will be maintained with Fi02 35%. Then, shortly before the planned extubation, Fi02 will be increased again to 80%.
  Interventions: Other: Oxygen

INTERVENTIONS:
Other: Oxygen — Delivery of high concentration of oxygen at induction, maintenance and extubation of children under general anesthesia.

SUMMARY:
This study is aiming at assessing the effect of inspired oxygen fraction during general anesthesia on children's lung mechanics and volume. More specifically, the temporal change in end-expiratory lung volume (EELV) and respiratory system resistance and elastance during the perioperative period will be characterized in order to define the the effect of high inspired fraction of oxygen on lung function.

DETAILED DESCRIPTION:
High-enriched oxygen fractions (FiO2)are common practice during general anesthesia both to ensure normoxemia despite intrapulmonary shunts and to provide security in case of adverse events. However, high-inspired oxygen fraction may decrease ventilation-perfusion ratios and its benefits are still unproven in children.

The investigators aim at assessing the benefits and potential adverse effects of high-inspired oxygen fraction in two groups of children receiving either 30% FiO2 or 80% FiO2 during maintenance of anesthesia. Nitrogen multiple breath washout technique and forced oscillation technique will be used to measure end-expiratory lung volume (EELV) and airway resistance (Rrs) and respiratory elastance (Xrs) respectively. These measurements will be obtained before the general anesthesia, one hour and one day after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) physical status I and II
* Body mass index < 30 kg/m2
* Scheduled for elective surgery in the supine position lasting < 200 min
* General Anesthesia with tracheal intubation

Exclusion Criteria:

* Patients hospitalized more than 24 h before the operation
* History or clinical signs of heart or lung disease
* Upper respiratory tract infection < 2 weeks prior to surgery
* Predictable difficult airway
* History of apnea
* Abdominal or thoracic surgery
* Lack of cooperation, language barrier

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2015-05; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Postoperative changes in lung volume in children receiving low (35%) or high (80%) intraoperative fraction of oxygen | 24 hours
  Measurement of end-expiratory lung volume by nitrogen wash-out technique
Postoperative changes in airway resistance in children receiving low (35%) or high (80%) intraoperative fraction of oxygen | 24 hours
  Measurement of airway resistance and respiratory system elastance by forced oscillation technique

SECONDARY OUTCOMES:
Respiratory complications | 1 month
  Assessing intraoperative (bronchospasm, laryngospasm, oxygen desaturation, airway obstruction) and postoperative (hypoxemia, atelectasis, pneumonia) complications
Postoperative nausea and vomiting | 24 hours

OTHER OUTCOMES:
Surgical site infection | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Walid Habre, MD, PhD, Study Director — Geneva Children's Hospital, University Hospitals of Geneva; Beatrice de la Grandville, Principal Investigator — Geneva Children's Hospital, University Hospitals of Geneva; Sam Bayat, MD, Principal Investigator — University Hospitals of Geneva
Locations (1):
- Geneva Children's Hospital, Pediatric Anesthesia Unit, Geneva, Switzerland

REFERENCES:
- [Derived] Grandville B, Petak F, Albu G, Bayat S, Pichon I, Habre W. High inspired oxygen fraction impairs lung volume and ventilation heterogeneity in healthy children: a double-blind randomised controlled trial. Br J Anaesth. 2019 May;122(5):682-691. doi: 10.1016/j.bja.2019.01.036. Epub 2019 Mar 11. PMID 30916028